CLINICAL TRIAL: NCT06912594
Title: Pilot Study to Investigate the Influence of an App on the Quality of Life and Symptoms of Patients With Polycystic Ovary Syndrome
Brief Title: App Impact on Quality of Life and Symptoms in PCOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endo Health GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: RCT_PilotPCOS
Record Dates: First submitted 2025-03-26; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: PCOS; Quality of Life; Digital Therapeutics
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Control group has access to care-as-usual only.
- Intervention Group (Experimental): The intervention group has access to the PCOS app and its functions in in addition to care-as-usual
  Interventions: Device: PCOS-App

INTERVENTIONS:
Device: PCOS-App — The PCOS-App helps to implement multimodal self-help measures in the daily lives of PCOS patients through various functions such as symptom diary and interactive exercises.
  Arms: Intervention Group

SUMMARY:
This study investigates the influence of a PCOS app on the quality of life and symptoms of individuals with polycystic ovary syndrome (PCOS). The intervention group can use the app over the study period of twelve weeks in addition to care-as-usual (CAU). In the control group, this is compared with no use of the PCOS-App for a twelve-week period, that is, care-as-usual only/ continuation of the current treatment (waitlist design). The aim is to evaluate the effectiveness of the app and to gain insights for the design of future studies. The study is expected to last seven months and include 220 participants.

DETAILED DESCRIPTION:
The study aims to investigate the effect of a PCOS app on quality of life and symptoms of individuals with polycystic ovary syndrome (PCOS). PCOS is a widespread and distressing health problem that can significantly affect quality of life and well-being of affected individuals. Research into digital health applications has shown the potential to provide innovative solutions to improve care and self-management of chronic conditions.

The present study is designed as a single-blind, two-arm, randomised controlled trial in which participants will either receive the PCOS app over a 12-week period in addition to care-as-usual (intervention group) or only care-as-usual as typically available (control group). The study will be conducted online. The aim is to evaluate the effectiveness of the app by analysing various questionnaires as endpoints. The primary endpoint is the Polycystic Ovary Syndrome Questionnaire (PCOSQ-G). The questionnaires/endpoints will be completed at T0 (baseline) and after 12 weeks. Statistical analyses will be conducted using R and SPSS. Exploratory evaluations of change scores in the relevant questionnaires will be performed.

Overall, this study aims to provide important insights into whether and to what extent a PCOS app can have a positive impact on the quality of life and symptoms of women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Legal capacity
* Resident in Germany
* Female gender
* Age ≥18 years up to 65 years
* Diagnosed and medically confirmed Polycystic Ovary Syndrome (E28.2)
* Ownership of a smartphone with a compatible iOS or Android version and the ability to operate it
* Internet access and an email address for registration, app usage, and completing questionnaires
* Willingness to complete questionnaires online
* Motivation to use the app regularly
* Sufficient knowledge of the German language

Exclusion Criteria:

* Changes in hormone therapy within eight weeks prior to the start of the study and/or planned within the next 12 weeks
* Changes in treatment with metformin within eight weeks prior to the start of the study and/or planned within the next 12 weeks
* Current treatment with medications for obesity (e.g., liraglutide, orlistat)
* Changes in treatment with anti-androgens (e.g., spironolactone, cyproterone acetate, flutamide) within eight weeks prior to the start of the study and/or planned within the next 12 weeks
* Pregnancy or breastfeeding
* Current hormonal fertility treatment
* Changes in treatment with psychotropic medications within eight weeks prior to the start of the study and/or planned within the next 12 weeks
* Current psychotherapeutic treatment
* Previous or current access to the Endo-App or other digital health applications (DiGAs)
* Current participation in other clinical studies
* Current nutritional counseling according to §20 SGB V or nutritional therapy according to §43 SGB V, or participation in weight reduction programs

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-04-02 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Polycystic Ovary Syndrome Questionnaire (PCOSQ-G) | From enrollment to the end of treatment at 12 weeks

SECONDARY OUTCOMES:
Body Appreciation Scale - 2 (BAS-2) | From enrollment to the end of treatment at 12 weeks
Patient Activation Measure 13 (PAM-13) | From enrollment to the end of treatment at 12 weeks
Depression Anxiety Stress Scale 21 Items (DASS-21) | From enrollment to the end of treatment at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Endo Health GmbH, Chemnitz, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No